CLINICAL TRIAL: NCT02663713
Title: A Randomized, Pharmacodynamic Comparison of Low Dose Ticagrelor to Clopidogrel in Patients With Prior Myocardial Infarction
Acronym: ALTIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Patras (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Dimitrios Alexopoulos, Professor, University of Patras
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: D5130C05274
Record Dates: First submitted 2016-01-21; First posted 2016-01-26 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Myocardial Infarction; Diabetes Mellitus; Renal Disease; Coronary Artery Disease
Keywords: Pharmacodynamics; Ticagrelor; Clopidogrel; MI
MeSH Terms: conditions — Myocardial Infarction; Diabetes Mellitus; Kidney Diseases; Coronary Artery Disease | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor (Experimental): Ticagrelor 60 mg twice daily
  Interventions: Drug: Ticagrelor; Drug: Clopidogrel
- Clopidogrel (Active Comparator): Clopidogrel 75 mg once daily
  Interventions: Drug: Ticagrelor; Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — Ticagrelor 60mg twice daily
Drug: Clopidogrel — Clopidogrel 75 mg once daily

SUMMARY:
Taken together the results from CHARISMA and PEGASUS-TIMI54, it appears that physicians may consider extending beyond 1 year or reinitiating treatment with clopidogrel 75 mg od or ticagrelor 60mg bid in patients with a prior MI and features of high ischemic and low bleeding risk. Comparative clinical or pharmacodynamic studies, however, between clopidogrel 75 mg od and ticagrelor 60 mg bid in the chronic phase of stable post MI patients have not been performed.

In a platelet substudy of PEGASUS-TIMI 54, 180 patients who had received >4 weeks of study medication had platelet reactivity assessment. Ticagrelor 60mg bid achieved high levels of peak and trough platelet inhibition in nearly all patients, with similar consistency of effect compared to 90mg bid. Platelet reactivity (PRU) was significantly reduced with ticagrelor 60mg bid compared to placebo.

In light of this, we believe that a dedicated pharmacodynamic study of ticagrelor 60 bid mg vs clopidogrel 75 mg od in a PEGASUS-like population would be informative for the practicing clinician, thus setting the rationale for conducting this specifically designed investigation.

This is a prospective, randomized, single blind, single center, crossover study. Eligible patients undergoing P2Y12 receptor antagonist therapy before screening will undergo a 14-day minimum washout period before randomization. Following screening/washout period (visit 1), patients will be randomized (visit 2, time 0) in 1:1 fashion to either clopidogrel 75 mg od or ticagrelor 60 mg bid. Following 14±2 days (visit 3) patients will receive alternate treatment for additional 14 days (visit 4). Platelet reactivity assessment will be performed with the VerifyNow P2Y12 reaction assay at time 0, prior to first study drug dose. At visit 3 platelet function will be assessed at 2-4 hours post dose and prior to crossover. At visit 4 also platelet function will be assessed at 2-4 hours post study drug post dose. All patients will receive concomitant aspirin (100 mg/d) and standard secondary prevention medication.

The primary endpoint is the platelet reactivity measured in P2Y12 reaction units (PRU) at the end of the 2 study periods (pre-crossover and post-crossover).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Post-menopausal female (defined as absence of any vaginal bleeding for a year) or male aged >50 years
3. A spontaneous MI (ST or Non ST segment elevation) 1 to 3 years before enrolment. In addition, at least one of the following high-risk features: age of 65 years or older, diabetes mellitus requiring medication, a second prior spontaneous MI, multivessel coronary artery disease, or non-end stage renal disease (estimated creatinine clearance of <60 ml per minute).

Exclusion Criteria:

1. Planned use of a P2Y12 receptor antagonist, dipyridamole, cilostazol, or anticoagulant therapy during the study period;
2. Known allergy, intolerance, hypersensitivity to ticagrelor or clopidogrel or any excipients,
3. Active pathological bleeding, severe hepatic impairment, a bleeding disorder or a history of an ischemic stroke or intracranial bleeding, a central nervous system tumor, or an intracranial vascular abnormality;
4. Gastrointestinal bleeding within the previous 6 months or major surgery within the previous 30 days;
5. Concomitant use of potent Cytochrome P450 3A4 (CYP3A4) inhibitors (atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin and voriconazole, grapefruit juice over 1 litre daily), CYP3A substrates with narrow therapeutic indices (cyclosporine, quinidine), or inducers (carbamazepine, dexamethasone, phenobarbital, phenytoin, rifampin, and rifapentine).
6. Increased risk of bradycardic events (e.g. known sick sinus syndrome or third degree AV block or previous documented syncope suspected to be due to bradycardia unless treated with a pacemaker).
7. Inability to adhere to the follow-up requirements or any other reason or condition that the investigator feels would place the patient at increased risk if the investigational therapy is initiated.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
platelet reactivity measured in P2Y12 reaction units (PRU) at the end of the 2 study periods (pre-crossover and post-crossover). | 14 days

SECONDARY OUTCOMES:
• High platelet reactivity rate (defined as >208 PRU) at the end of the 2 study periods | 14 days
• VerifyNow P2Y12 assay % inhibition, using the TRAP-induced (BASE channel) response at the end of the 2 study periods | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology Department Patras University Hospital, Rio, Achaia, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730